CLINICAL TRIAL: NCT04842851
Title: Cardiac Resynchronization Therapy in Congenital Heart Diseases With Systemic Right Ventricle
Status: Completed | Type: Observational
Sponsor: Paris Cardiovascular Research Center (Inserm U970) (Other Government)
Collaborators: Marie Lannelongue Hospital, Le Plessis Robinson, France (Unknown); Clinique Pasteur Toulouse (Other); Groupe Hospitalier Pitie-Salpetriere (Other); Hopital Louis Pradel (Other); University Hospital, Montpellier (Other); European Georges Pompidou Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2219047
Record Dates: First submitted 2021-04-06; First posted 2021-04-13 (Actual); Last update posted 2021-04-13 (Actual); Status verified 2021-04

CONDITIONS: Congenital Heart Disease
Keywords: cardiac resynchronization therapy; congenital heart disease; systemic right ventricle; outcomes
MeSH Terms: conditions — Heart Defects, Congenital | interventions — Cardiac Resynchronization Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: cardiac resynchronization therapy — Cardiac resynchronization therapy in patients with systemic right ventricle

SUMMARY:
This study aims to analyze outcomes of patients with systemic right ventricle (SRV) implanted with Cardiac Resynchronization Therapy (CRT) systems and to compare the impact of CRT in SRV patients with other congenital heart diseases (CHD).

DETAILED DESCRIPTION:
Heart failure is henceforth the main cause of death in adult patients with congenital heart disease (CHD). The number of affected patients is expected to continue to grow exponentially due to the important increase and aging of this population.

In symptomatic patients despite optimal pharmacological therapy, Cardiac Resynchronization Therapy (CRT) offers a well-recognized therapeutic option in dilated and ischemic cardiomyopathies with severely impaired left ventricle ejection fraction and complete left bundle branch block. In patients with CHD, the level of evidence is much more limited. Underlying phenotypes are heterogeneous, including systemic right ventricles (SRVs), isolated sub-pulmonary right ventricle dysfunctions, single ventricles, and most of patients have a right bundle branch block. All these specificities question the extrapolation of data reported in patients with acquired cardiomyopathies. Despite the lack of evidence, CRT systems have been progressively used in CHD patients, also because alternative options are poor, mainly represented by cardiac transplantation, but grafts are rare and congenital patients frequently have contraindications.

A positive impact of CRT in CHD has first been suggested in small series where hemodynamic invasive parameters (e.g. dP/dt max) were improved and QRS narrowed by multisite pacing. A few subsequent studies then reported an improvement of ventricular functions and patient-reported functional subjective parameters (mainly NYHA classification). However, the number of patients included in most studies was limited and heterogeneous forms of CHD were often pooled when interpreting results. The studies evaluating CRT specifically in patients with SRV are very rare and demonstrated conflicting results. The largest study to date assessing specifically CRT in patients with SRV included 20 patients with congenitally corrected transposition of the great arteries (cc-TGA) and demonstrated an acute improvement in two-thirds of patients.

Although patients with SRV represent one of the main groups of CHD patients currently implanted with CRT, the paucity of specific data in this population has been highlighted as a major evidence gap and as a high-impact research question by the American Heart Association/American College of Cardiology guidelines committee.

ELIGIBILITY:
Inclusion Criteria:

* All patients with congenital heart disease and CRT device

Exclusion Criteria:

* Patient's refusal

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients with congenital heart disease and CRT device. The group of patients with systemic right ventricle include patients with D-transposition of the great arteries (D-TGA) with atrial switch operation (Mustard or Senning surgery) and patients with congenitally-corrected transposition of the great arteries (cc-TGA) with SRV (excluding cc-TGA with systemic left ventricle post surgical repair, e.g., arterial switch procedure or Rastelli surgery).
Sampling Method: Probability Sample
Enrollment: 85 (Actual)
Dates: Start 2004-01-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with response to CRT | 6-month, 12-month, 24-month
  Proportion of patients with improvement of NYHA classification by at least one grade or improvement of systemic ventricular ejection fraction by at least 10%
Proportion of patients with response to CRT | 12-month
  Proportion of patients with improvement of NYHA classification by at least one grade or improvement of systemic ventricular ejection fraction by at least 10%
Proportion of patients with response to CRT | 24-month
  Proportion of patients with improvement of NYHA classification by at least one grade or improvement of systemic ventricular ejection fraction by at least 10%

SECONDARY OUTCOMES:
Overall mortality | 5 and 10 years
  All cause mortality
Overall mortality or heart transplantation | 5 and 10 years
  All cause mortality or heart transplantation
Complications associated with CRT | Acute (<30 days after procedure) and late (>30 days)

CONTACTS AND LOCATIONS:
Overall Officials: Victor Waldmann, MD, PhD, Principal Investigator — Georges Pompidou European Hospital, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided